CLINICAL TRIAL: NCT03330340
Title: Percutaneous Vertebroplasty Versus Conservative Treatment in Vertebral Compression Fracture Associated With Glucocorticoids-induced Osteoporosis: a Prospective Cohort Study
Brief Title: Percutaneous Vertebroplasty Versus Conservative Treatment in GIOPVCF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Haolin Sun, Clinical Professor, Peking University First Hospital
Other Study IDs: HSun-1
Record Dates: First submitted 2017-10-08; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Osteoporosis
Keywords: vertebral compression fracture; osteoporosis; glucocorticoids; vertebroplasty
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Percutaneous vertebroplasty: All PVPs are performed by experienced spine surgeons under optimal fluoroscopic guidance. The procedure takes place under sterile conditions. Local anesthesia is administered to the periosteum of the targeted pedicle via skin. Polymethylmethacrylate bone cement is injected under continuous fluoroscopic guidance using 1.0 ml syringes and 13 Gauge bone biopsy needles by bilateral procedures. Patients are encouraged to stand up and walk with brace immediately after operation and the brace are required to be worn for 3 months. Furthermore, all patients will take oral bisphosphonates treatment together with supplemental calcium and vitamin D.
  Interventions: Procedure: Percutaneous Vertebroplasty
- Conservative treatment: In conservative treatment group, the patients were required horizontal bed rest for the initial 2 weeks after diagnosis. Then, they were encouraged to stand up and walk with brace and assistance. The bed rest time was extended if the back pain worsened when they stood up and walked. The brace should be worn in 3 months. For pain medication, nonsteroidal anti-inflammatory drugs (NSAIDs) were prescribed for every patient. Additional analgesics, such as tramadol and morphine, would be added in case NSAIDs were not effective. Two weeks after diagnosis, physical therapy was started. All patients are put on osteoporosis medication, bisphosphonates together with supplemental calcium and vitamin D.

INTERVENTIONS:
Procedure: Percutaneous Vertebroplasty — The procedure takes place under sterile conditions. Local anesthesia is administered from skin to the periosteum of the targeted pedicle. Polymethylmethacrylate bone cement (Mendec Spine; Tecres SPA, Sommacampagna, Italy) is injected under continuous fluoroscopic imaging guidance using 1.0 ml syringes and 13 Gauge bone biopsy needles by bilateral procedures. The amount of injected cement in each treated vertebral body and any cement leakage is recorded.
  Groups: Percutaneous vertebroplasty

SUMMARY:
Based on the case reports and other literature, the investigators hypothesize that using PVP for treating GIOPVCF is associated with increased risk of vertebral refractures and does not provide further benefits compared to conservative treatments.

The overall objective of this prospective cohort study is to compare the efficacy of PVP and conservative treatment for GIOPVCF. The evaluation of efficacy of therapy includes: 1) the incidence of vertebral refractures; 2) therapeutic effects (pain relief and health-related life quality) and 3) complications.

The results from study will be written in English and disseminated widely through scholarly presentations, peer-reviewed publications, and other written communications.

DETAILED DESCRIPTION:
Patient recruitment and informed consent The study will recruit patients with GIOPVCF after consultation with inpatients and outpatients. The principal investigator of the study will screen the clinical information and inform the patients whether they are eligible for the study. After explaining the two therapeutic strategies (conservative treatment and PVP) and signing the informed consent, the patients will be divided into conservative treatment or PVP group based on their own decision.

The general information and medicine history of the participants are collected: age, gender, original disease, the course of original disease, specific GCs that have been used, the dosage/length of the GCs treatment, specific anti-osteoporosis medicine have been used and the dosage and length of usage. The bone density of the patient will then be evaluated using Dual-energy X-ray absorptiometry (DXA).

Withdrawal of individual subject Patients can withdraw from the study at any time for any reason without any consequences. The investigator can also decide to release patients from the study for medical reasons. For every patient who decides to withdraw from the study, the reasons of withdrawal will be recorded.

Sample size calculation A p-value is less than significance level (α) of 0.05 is considered as statistically significant. The statistical power (1-β) is defined as 80%. Based on the survival analysis of primary endpoint , the incidence of refracture in the patients with GIOPVCF is 48.6% after initial PVP operation and 17% after initial conservative treatment. Thus, power analysis indicates the study requires 42 patients per group to achieve statistical significance between two groups. Considering 20% of patients may be lost during follow-up visits, the investigators will recruit 53 patients for each group.

Statistical analysis Standard statistical techniques will be used to describe characteristics of patients in both groups. The investigators will compare baseline characteristics in the two treatment groups and if incomparability appears, the investigators will in secondary analysis adjust for differences. The incidence of vertebral refracture between groups will be compared with the Kaplan Meier survival analysis. Baseline differences of pain relief and health-related life quality between two groups will be assessed using student t test or nonparametric tests. Changes of VAS, ODI, and EQ-5D within the group from baseline to every follow-up time point will be compared using paired t test. A P value less than 0.05 is considered as statistically significant. SPSS 17.0 statistical program (SPSS, Chicago, IL) will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have fresh vertebral compression fractures regarding spine radiograph (minimum 15% height loss; level of fracture at Th5 or lower; bone edema on MRI, focal tenderness on VCF level).
2. Patients have back pain for 6 weeks or less, with a visual analogue scale (VAS) score equal or less than 5.
3. GCs consumption for more than 3 months (prednisone equivalent or more than 5 mg daily).
4. Reduced bone density with T-scores equal or less than -1.
5. Age at 55 or higher.

   -

Exclusion Criteria:

1. Concurrent other secondary osteoporosis.
2. Previous PVP procedure or other spinal surgery on thoracic or lumbar segments.
3. Systemic or local infection in spine (osteomyelitis, spondylodiscitis)
4. Unable to comply with study due to severe psychosis.

   -

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had fresh vertebral compression fractures with GIOP
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of vertebral re-fracture | 12 months after the treatment
  Anterior-posterior and lateral spinal radiograph will be obtained. If a new vertebral fracture was doubted, MRI was undertaken to confirm it. When there is disagreement between both observers a consensus meeting is held. Incidence of vertebral re-fracture is Number of new fracture vertebrae/Number of total vertebrae

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for back pain change from baseline to 12 months | 12 months after the treatment
  All participants are asked to fill out standard questionnaires of the VAS score for back pain. The VAS pain is a single-item scale. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10). The change from baseline to 12-month post treatment will be compared between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Li, Doctor, Study Director — Peking University First Hospital